CLINICAL TRIAL: NCT00880802
Title: Finding ACS With Serial Troponin Testing for Rapid Assessment of Cardiac Ischemic Symptoms
Brief Title: Finding Acute Coronary Syndromes (ACS) With Serial Troponin Testing for Rapid Assessment of Cardiac Ischemic Symptoms
Acronym: FAST-TRAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanosphere, Inc. (Industry)
Responsible Party: Greg Shipp, MD / Chief Medical Officer; VP, Medical and Regulatory Affairs, Nanosphere, Inc.
Other Study IDs: FAST-TRAC
Record Dates: First submitted 2009-04-11; First posted 2009-04-14 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Non ST-Segment Elevation Myocardial Infarction; ST-Segment Elevation Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Objectives

The following items will be prospectively assessed.

Primary Endpoints

1. For patients presenting with clinical suspicion of Acute Coronary Syndromes (ACS), high sensitivity-cardiac Troponin I (hs-cTnI) provides improved diagnostic accuracy for ACS (including Acute Myocardial Infarction (AMI) and/or Unstable Angina (UA)) within the first two (2) hours after emergency department presentation when compared to currently available troponin assays.
2. For patients presenting with clinical suspicion of ACS, hs-cTnI provides improved prognostic information with regard to 180 day event rates of Major Adverse Cardiac Event outcomes, including cardiac deaths which are defined as all deaths except those that are clearly non-cardiac in nature (e.g. trauma), when compared to a currently available troponin assay.

Secondary Endpoints

1. For patients presenting with clinical suspicion of ACS, using the rate of rise of hs-cTnI over time between presentation and 2 hours (delta hs-cTnI) allows for the differentiation between ACS and other disease states.
2. For patients presenting with clinical suspicion of ACS, hs-cTnI provides improved sensitivity for detecting AMI within the first two (2) hours after presentation when compared to a currently available troponin assay.
3. For patients presenting with clinical suspicion of ACS, hs-cTnI provides improved negative predictive value for ruling out ACS (AMI or UA) within the first 2 hours after presentation when compared to a currently available troponin assay.
4. For alternative endpoints of cardiac mortality, and for alternative censor time points of 30 days, 90 days, and 1 year, hs-cTnI provides improved prognostic information when compared to the currently available troponin assay.
5. In cases where the emergency physician has limited diagnostic confidence, hs-cTnI AMI diagnostic accuracy will be superior to local hospital standards for AMI determination.
6. In cases where the emergency physician has limited diagnostic confidence, the slope for the hs-cTnI between presentation and 2 hours will add diagnostic accuracy for ACS diagnosis over and above local hospital standards for ACS determination.
7. For patients presenting with clinical suspicion of ACS, the difference in diagnostic accuracy for ACS (including AMI and/or UA) using hs-cTnI measurement from time of onset of symptoms to emergency department presentation (e.g. 3 hours instead of 6 hours) will be evaluated to assess any variation.

DETAILED DESCRIPTION:
This study will evaluate the ability of a high sensitivity cardiac troponin I (hs-cTnI) assay to detect and to rule-out high-risk ischemic cardiac injury in emergency room patients experiencing signs and symptoms consistent with acute coronary syndromes (ACS). Cardiovascular disease is still the most frequent cause of morbidity and mortality among industrialized nations. In the U.S., there are nearly 100 million adults who suffer from cardiovascular disease. Over 5 million patients present to emergency departments (EDs) annually with a chief complaint consistent with ACS. A majority of these patients are found to be experiencing non-cardiac chest pain (about 70-82% of patients). Myocardial infarction (MI, including non-ST-segment elevation MI [NSTEMIs = about 6-10% of patients] and ST-segment elevation MI [STEMIs = about 2-5% of patients]) occurs in about 8-15% of these patients. Unstable angina (UA), which is often a precursor condition to MI, accounts for 10-15% of patients. Together, MI plus UA combine to define ACS (= about 18-30% patients).

MI is caused by rupture of an atherosclerotic plaque in a coronary artery, leading to platelet aggregation and thrombus formation to an extent that oxygenation of the myocardial tissue is completely interrupted (i.e., total occlusion), with the occurrence of some degree of myocardial necrosis. High concentrations of cardiac enzymes and proteins (e.g., cardiac troponin I or T [cTnI or cTnT], CK-MB, myoglobin) are observed in blood as the result of significant irreversible injury to cardiac tissue distal to the site of rupture and secondary to arterial occlusion. Current assays can detect STEMIs and NSTEMIs but, by definition of the 2007 AHA/ACC updated guidelines for NSTEMI and UA, the NSTEMI threshold is defined as the 99th percentile upper reference limit [URL] of a cardiac troponin (cTn) assay's reference range in a healthy subject population, and they cannot detect what is currently labeled "unstable angina (UA)" or ischemia without necrosis. In addition, it typically takes 4-6 hours, after ischemic symptoms begin, for the cardiac troponin to rise above the current commercial assay NSTEMI threshold (i.e., the upper reference limit [URL] = the 99th percentile upper reference limit). These issues expose a sensitivity problem with current generation cTn assays, including the most sensitive tests available.

UA is also associated with plaque rupture but only partial coronary artery occlusion occurs, resulting in ischemic pain but no (or unmeasureable) necrosis. No rise is observable in cardiac marker levels on currently available assays (best limit of detection [LOD] of ~0.01 ng/mL [10 pg/mL] and best URL of ~0.03 ng/mL [30 pg/mL]). Since there is no test currently available that accurately diagnoses UA, many UA patients are discharged home in the midst of a high-risk ischemic event. (Note: Ischemia modified albumin [IMA] is on the market but is not widely used due to its poor specificity.) The negative predictive value of the diagnostic test is important in this regard, as increases in sensitivity may be offset if there are also increases in false positive results.

As many as 2% (30,000 patients) to 4% (60,000 pts) of patients with MI or UA (~750,000 MI patients + ~750,000 UA patients = ~1.5 million total patients at risk) are inadvertently discharged from the ED with an associated short-term mortality of 10% to 26% (Duseja and Feldman 2004). Missed acute cardiac ischemia is one of the major causes of malpractice litigation against emergency physicians (Duseja and Feldman 2004). Even though chest pain (and other symptoms consistent with ACS) patients represent only 6% of the ED patient volume, it has been estimated that 20% of ED-related malpractice dollars are expended for ischemic heart disease complications (Rusnak, et al 1989). Therefore, the misdiagnosis of ischemic cardiac injury is of great importance from a human-life and economic perspective.

In the typical hospital ED today, cardiac biomarkers are drawn and the results are back to the ED physician within about 1.5 hours (i.e., therapeutic turnaround time [TTAT]; "vein to brain" time). Some hospitals have moved to point-of-care devices (with relatively low sensitivity [URL = 0.080 ng/mL]) that can give results within 10-15 minutes and, on the other extreme, some EDs that are still dependent on the central laboratory have a therapeutic turnaround time of 2-4 hours. Most chest pain patients that continue to have discomfort and other cardiac symptoms are held in the ED or chest pain (observation) unit for 6 to 23 hours, before discharge, allowing serial cardiac markers to be drawn. Therefore, keeping these time points in mind, a highly sensitive (e.g., URL = 0.003 ng/mL) and precise cTn assay (e.g., <20-30%CV) that takes < 1 hour to give a result may be very useful for any hospital ED.

Time is important but, in the case of ischemic heart disease, accurate information is more important and is potentially life-saving. The information that the assay would give to the ED physician would allow for accurate diagnosis of what is currently labeled "UA" and not discharge a patient who actually requires close monitoring, treatment, or follow-up at a cardiologist's office. Also, the diagnosis of an MI could be made much earlier (with high sensitivity and specificity) than the 4-6 hours after ED presentation that it takes for cTn to be detected by current assays.

With no cardiac marker assay available that can diagnose "UA" with appropriate accuracy and precision, development of a cost-effective, timely (< 1 hr assay time) cardiac troponin assay that allows accurate measurement of cTn at concentrations that are 10-100 fold below the best of the current assays' detection limits has the potential to improve ACS patient care. It will allow diagnosis of ischemic injury in "UA" patients in the ED so they can be admitted appropriately to the hospital instead of being sent home to experience a possible cardiac event or death. With current therapeutic capabilities (e.g., LMWHs, beta-blockers, glycoprotein IIb/IIIa inhibitors, other anti-platelet agents) that are known to lower the risk of future cardiac events and mortality, it can be expected that the earlier detection of MI and diagnosis of "UA" may lead to reductions in morbidity and mortality in ACS patients.

The need for a highly sensitive assay for cardiac troponin is predicated on the observation that the URL of the true reference range in nominally healthy subjects is significantly below the concentrations that current assays can measure. A new nanoparticle-based, highly sensitive cTnI assay (i.e., nano-assay) appears to offer a significant technological advantage over the current macroparticle-based, sensitive assays. The new highly sensitive assay's LOD is ~800 fg/mL (800 fg/mL = 0.8 pg/mL = 0.0008 ng/mL) for cardiac troponin I, as compared to 10 pg/mL (0.010 ng/mL) for the most sensitive cTnI assay currently on the market. The new assay has an imprecision (%CV), at the LOD, of <20-30%, as compared to >>30% at the LOD for the most sensitive cTnI assay currently on the market. The URL of the reference range in healthy subjects for the new assay is about 2.8 pg/mL (0.0028 ng/mL), compared to 30 pg/mL (0.030 ng/mL) for the most sensitive cTnI assay currently on the market. Under these differences in analytical performance, it is likely that the majority of patients with what is currently labeled "UA" will reveal detectable troponin concentrations that exceed the nano-assay's threshold limit (i.e., 2.8 pg/mL = 0.0028 ng/mL) on the nanoparticle-based, highly sensitive cTnI assay but non-detectable levels of troponin on the current macroparticle-based, sensitive cTnI assays.

In a pilot study, banked serial serum samples of ten NSTEMI patients from the Hospital of the University of Pennsylvania ED were evaluated on a research version of the nano-assay. These serial samples were "troponin-negative" on an older laboratory assay (laboratory assay URL = 0.6 ng/mL = 600pg/mL) for the first 1-3 blood draws. Samples from these patients at presentation, 90min, and 180min were measured by a current sensitive assay (Siemens [Dade Behring] Stratus CS) sensitive assay URL = 0.070ng/mL = 70pg/mL) and by the experimental highly sensitive assay (highly sensitive assay URL=0.0028 ng/mL = 2.8 pg/mL). None (0%), two (20%), and ten (100%) of the ten NSTEMI patients were found to be cTnI positive at presentation on the laboratory, sensitive, and highly sensitive assays, respectively. All 10 patients measured at >35pg/mL on the highly sensitive assay at presentation. Three of the patients remained "cTnI negative" for >180 min on the current sensitive assay.

In another research study, samples from 100 chest pain patients with known ACS (i.e., 50 NSTEMI and 50 "UA" patients) were evaluated. Comparison was made between the laboratory device and the highly sensitive nano-assay with a URL of 0.0028 ng/mL (2.8 pg/mL). Using the current laboratory assay (Siemens [Dade Behring] Dimension; URL = 0.100 ng/mL = 100 pg/mL), the 50 NSTEMI patients were cTnI negative on the first draw, and the 50 "UA" patients were cTnI negative throughout their stay in the ED and/or hospital. At presentation (t = 0 hrs), 7 hrs, and 24 hrs, none (0%) of the "UA" patients were found to be positive for cTnI on the laboratory instrument. Using the nano-assay with the same "UA" patients' serum samples, 48%, 64%, and 82% were positive for cTnI at presentation, 2 hrs, and 7 hrs, respectively. For the NSTEMI patients at presentation (t = 0 hrs), 7 hrs, and 24 hrs, none (0%), 56%, and 98%, respectively, of the patients were found to be positive for cTnI on the laboratory instrument. Using the nano-assay with the same NSTEMI patients' serum, 76%, 98%, and 100% were positive for cTnI at presentation, 2 hrs, and 7 hrs, respectively.

These preliminary results demonstrate the potential strength of this highly sensitive cTnI assay to reveal an abnormal [cTnI] at ED presentation that may progress to MI (i.e., NSTEMI or STEMI) and to detect acute ischemic insult that may not progress to MI (i.e., "UA"). This high sensitivity protein assay may enhance the clinical utility of testing for ACS in the ED and other cardiac care settings (e.g., earlier detection leading to directed therapies, improve risk stratification, earlier rule-out of non-cardiac-related chest pain [NCCP], detection of re-infarction).

The definition of myocardial infarction used in this study will be the meaning that was recently updated and published in the November 27, 2007 issue of Circulation (Thygesen, et al 2007). Page 18 of this study protocol contains this definition. The definition is based on cardiac troponin as the biomarker of choice with any value above the 99th percentile of an assay's reference range population considered abnormal. Therefore, if the nano-assay's URL is much lower than the current assay's URL, all values that are above the nano-assay's URL but below the current assay's URL that were considered "UA" on the current assay should now be considered myocardial infarction when measured on the nano-assay. This may result in the "UA" category being removed as an ACS categorization.

There are also recent studies (Zethelius, et al 2006; Waxman, et al 2006) that show very low cTnI values (<30-40 pg/mL) can predict future cardiac events and mortality in the asymptomatic elderly male population (>70 years) and in symptomatic ED patients with cTnI levels that remain in the reference (normal) ranges of current assays. A highly sensitive assay that could detect "silent" cardiac damage in these cTnI ranges in the cardiologist's office and ED settings could be a predictor of future risk that could direct appropriate therapeutics and preventative care.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age or older.
* The subject must present to the Emergency Department with symptoms consistent with acute coronary syndromes (e.g., chest discomfort/pain, squeezing/fullness in the chest, pain radiating to left or both arms, jaw pain, pain in back/neck/stomach, shortness of breath, cold sweat, nausea/vomiting, lightheadedness).
* The subject must present to the Emergency Department within six (6) hours of the onset of the most recent symptoms that prompted the subject to seek medical attention in the Emergency Department.
* The subject agrees to abide by the protocol, including all telephone follow-up.

Exclusion Criteria:

* The subject is in acute distress and requires immediate life-saving intervention.
* The subject has experienced CPR, defibrillation, or cardioversion within 24 hours of presentation to the Emergency Department.
* The subject cannot give consent or understand the informed consent form.
* The subject has a terminal illness (e.g. metastatic cancer) and is not expected to survive 6 months.
* Patient has trauma related ACS symptoms (i.e. penetrating wounds, crush injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to evaluate cTnI in heparinized plasma at more frequent intervals than most rapid rule-out or rule-in protocols from ED subjects who: 1) are experiencing signs and symptoms consistent with ACS or ischemic heart disease in the ED, 2) have their initial ECG analysis performed in the ED, and 3) are expected to have cTnI measured serially in the ED.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
All enrolled patients will have subject diagnosis (non-ACS, ACS [MI or UA]) assessed utilizing a "Gold Standard" adjudication process. Timing of ACS diagnosis (per cTnI level and change) by hs-cTnI and currently available cTnI assay will be compared. | 30 days after enrollment completion
All enrolled patients will be followed up at 30, 90 and 180 days, and 1 year. Outcome information that will be assessed includes mortality, cardiac re-hospitalization, cardiac events, and re-vascularization. | 30 days, 90 days, 180 days and 1 year after the primary incident

SECONDARY OUTCOMES:
Using the rate of rise of hs-cTnI over time between presentation and 2 hours (delta hs-cTnI), differentiation between ACS and other chronic disorders may be possible. | 30 days after enrollment completion
Measuring the hs-cTnI level at a given threshold, may provide improved negative predictive value for ruling-out ACS (AMI or UA) within the first 2 hours after presentation. | 30 days after enrollment completion

CONTACTS AND LOCATIONS:
Overall Officials: W. Frank Peacock, MD, Principal Investigator — The Cleveland Clinic; Christian Mueller, MD, Study Chair — University Hospital, Basel, Switzerland; Alan S Maisel, MD, Study Chair — Veterans Affairs Medical Center San Diego and University of California, San Diego
Locations (16):
- United States (13):
  - University of California, Davis, Davis, California
  - University of California San Diego, San Diego, California
  - Veterans Affairs Medical Center San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Joseph Hospital, Bellingham, Washington
- Unversity of Athens, Attikon, Athens, Greece
- Sant'Andrea Hospital, Rome, Italy
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Peacock WF, Maisel AS, Mueller C, Anker SD, Apple FS, Christenson RH, Collinson P, Daniels LB, Diercks DB, Somma SD, Filippatos G, Headden G, Hiestand B, Hollander JE, Kaski JC, Kosowsky JM, Nagurney JT, Nowak RM, Schreiber D, Vilke GM, Wayne MA, Than M. Finding acute coronary syndrome with serial troponin testing for rapid assessment of cardiac ischemic symptoms (FAST-TRAC): a study protocol. Clin Exp Emerg Med. 2022 Jun;9(2):140-145. doi: 10.15441/ceem.21.154. Epub 2022 Jun 30. PMID 35843615